CLINICAL TRIAL: NCT06758843
Title: A Prospective, Controlled, Parallel Trial of Comparing Relative Peripheral Refraction Between Parameters Before and After Myopia Progression with Multispectral Refraction Topography
Brief Title: Comparing Relative Peripheral Refraction on Myopia Progression
Acronym: CMPMRT
Status: Completed | Type: Observational
Sponsor: Fuzhou Southeast Institute of Visual Ophthalmology (Other)
Responsible Party: Sponsor
Other Study IDs: Ningbo Eye Hospital; 2020Y55 (Other Grant/Funding Number: the Science and Technology Program of Ningbo, China)
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: Myopia progression; Peripheral myopia defocus; children; Refraction
MeSH Terms: conditions — Myopia | interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — ocular axial length, visual acuity, refractive error, peripheral retina refraction parameters such as total MRT value of both eyes, 15 degree MRT value, 30 degree MRT value, 45 degree MRT values, superior MRT values, inferior MRT values, nasal MRT values, temporal MRT values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fast progression group of myopia: The axial length elongation is equal or larger than 0.40 mm per year
  Interventions: Other: measure the axial length, visual acuity, and refraction at follow-up of 6- and 12-month
- Slow progression group of myopia: The axial length elongation is less than 0.30 mm per year
  Interventions: Other: measure the axial length, visual acuity, and refraction at follow-up of 6- and 12-month

INTERVENTIONS:
Other: measure the axial length, visual acuity, and refraction at follow-up of 6- and 12-month — the intervention is follow-up with parameters to measure and data to record

SUMMARY:
The investigators will test our hypothesis that parameters on peripheral defocus can regulate eye growth: For instance, the relative peripheral refraction measured by Multispectral Refraction Topography (MRT) would be significant different between two groups: fast speed and slow speed of axial length elongation (myopia progression) for 1 year with 2-3 follow-ups.

The goal of this observation study is to confirm the value of MRT in clinic. Could it predict myopia progression or not? By the parameters on relative peripheral refraction in children myopia, could include any of the following: both genders, 7~17 years age groups, including healthy volunteers. The main question it aims to answer is:

Is any of relative peripheral refraction parameters measured by MRT could guide the clinics for predict myopia progression? Which parameters from MRT could predict the myopia fast progression at baseline ? There is a comparison between groups. Researchers will compare fast myopia progression group versus slow myopia progression group to see if any parameters differs at baseline.

Participants will be asked to the collection methods (such as spectacles, orhtokeratology, contact lens) and interventions; And each participant would be followed up for at least 2 times in one year to test the axial length and refractive error as well as parameters with MRT.

DETAILED DESCRIPTION:
Visual signals from the surrounding retina play a crucial role in the process of emmetropization in the peripheral area of retina and may be a key factor in the development of myopia.

Peripheral defocus can regulate eye growth, particularly peripheral hyperopic defocus, which is a high-risk factor for promoting eye growth and the onset and progression of myopia.

In recent years, with the establishment of new experimental animal models and the emergence of new detection technologies, the relationship between peripheral defocus and myopia has received increasing attention.

The axial length of the eye is the most important indicator for assessing myopia progression.

About 7000 students from Ningbo would be follow-up for the MRT and their myopia progression for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Will to attend the baseline and all the follow-ups
* Sign the Inform Consent Form
* Could co-operate to ask for the correction and accept the axial length measurement and refraction devices including MRT
* Without eye surgery and trauma history
* His/Her refractive error and axial length could be measured

Exclusion Criteria:

* Without data of primary outcome
* With only one measurement
* Others condition that investigators consider not elilgible

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children in primary school and middle school, heathy or myopia at baseline
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2022-07-23 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Total value of relative peripheral refraction from MRT (D) | 12 months
  The parameter obtained using MRT for analysis is = total peripheral refraction - central refractive error.
Total relative peripheral refraction from MRT (D) | 6 months
  The parameter obtained using MRT for analysis
  * total peripheral refraction error - central refractive error

SECONDARY OUTCOMES:
Superior peripheral myopic defocus (D) | 12 months
  which indicates the average peripheral refractive error from the center to the peripheral of superior area of the retina.
peripheral refraction difference value 15 degree (D) | 12 months
  which indicates the average paracentral refractive error from the center to 15◦ of the retina
Peripheral refraction difference value-30 (D) | 12 months
  which indicate the average peripheral refractive error at 30 ◦
refraction difference value- 45 which indicate the average peripheral refractive error at 45◦ of the posterior retina (D) | 12 months
  the relative refraction difference value- 45which indicate the average peripheral refractive error at 45◦ of the posterior retina measured by MRT
relative refraction difference value-inferior (D） | 12 months
  the relative refraction difference value of inferior, which is measured by MRT
relative refraction difference value-nasal (D) | 12 months
  the relative refraction difference value-nasal measured by MRT
relative refraction difference value-temporal (D). | 12 months
  the relative refraction difference value-temporal measured by MRT.
Change of refractive error (D) | 12 months
  the change of refractive error is measured by auto-refractor without cycloplegia
Visual acuity (decimal ) | 12 months
  the visual acuity is test with decimal visual acuity chart at distance
Visual acuity (decimal ) | 6 months
  the visual acuity is test with decimal visual acuity chart at distance
Superior peripheral myopic defocus (D) | 6 months
  which indicates the average peripheral refractive error from the center to the peripheral of superior area of the retina.
peripheral refraction difference value 15 degree (D) | 6 months
  which indicates the average paracentral refractive error from the center to 15◦ of the retina
Change of refractive error (D) | 6 months
  the change of refractive error is measured by auto-refractor without cycloplegia
relative refraction difference value-inferior (D） | 6 months
  the relative refraction difference value of inferior, which is measured by MRT
relative refraction difference value-nasal (D) | 6 months
  the relative refraction difference value-nasal measured by MRT
refraction difference value- 45 which indicate the average peripheral refractive error at 45◦ of the posterior retina (D) | 6 months
  the relative refraction difference value- 45which indicate the average peripheral refractive error at 45◦ of the posterior retina measured by MRT
Peripheral refraction difference value-30 (D) | 6 months
  which indicate the average peripheral refractive error at 30 ◦

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Eye Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No